CLINICAL TRIAL: NCT05723367
Title: Perfusion Index Value in Predicting the Clinical Outcome of Lumbar ESPB
Brief Title: Prediction of Clinical Outcome in Lumbar ESPB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2023-01-025-03
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lumbar ESPB group where ESPB is performed at L4 with local anesthetics 20ml — ultrasound guided fascial plane injection

SUMMARY:
The primary endpoint of this study was to identify that Perfusion index (PI) has any predictive value for the treatment outcome of cervical radiculopathy

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. Although the special probe for PI measurement is relatively more expensive compared with ordinary pulse oximetery probes, its benefit as a marker of peripheral perfusion and as an idex for sympathetic stimulation have increased its use progressively. PI has been used widely for the prediction of success of brachial plexus block or axillary block. Changes of PI ratio value showed an excellent predictive value for the success of block.

There have been no studies demonstrating predictive value of PI in lumbar ESPB ESPB for the relief of low back pain or leg pain due to lumbar disc herniation or stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar foraminal stenosis
* Lumbar central stenosis
* Lumbar disc herniation
* Lumbar spondylolisthesis

Exclusion Criteria:

* Infection
* Pregnancy
* allergy to local anesthetic agnets
* Previous lumbar spine surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit the pain clinic
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Perfusion index changes among 4 time periods | baseline, 10 minutes after erector spinae plane block, 20 minutes after erector spinae plane block, 30 minutes after erector spinae plane block
  Perfusion index changes among 4 time periods
Number of patients showing numerical rating scale reduction more than 50% | 1 month after erector spinae plane block
  Number of patients showing numerical rating scale reduction more than 50%
Number of patients showing numerical rating scale reduction less than 50% | 1 month after erector spinae plane block
  Number of patients showing numerical rating scale reduction less than 50%
Number of patients showing no reduction in numerical rating scale | 1 month after erector spinae plane block
  Number of patients showing no reduction in numerical rating scale
Back pain functional scale between 2 time periods | baseline, 1 month after erector spinae plane block
  Back pain functional scale between 2 time periods

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Hoon Park, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No